CLINICAL TRIAL: NCT00005336
Title: Dietary Treatment of Hyperlipidemia in Women vs. Men
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4195; R01HL044878 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypercholesterolemia

SUMMARY:
To conduct a dietary intervention trial to test the lipid lowering response to the National Cholesterol Education Program (NCEP) Step Two Diet by free-living hyperlipidemic women and men and to compare the response between them.

DETAILED DESCRIPTION:
BACKGROUND:

Women experience as much illness from hardening of the arteries including stroke and heart disease as do men, but because women experience them later in life, the importance of heart disease, cholesterol, and diet for women has been under appreciated.

DESIGN NARRATIVE:

Half of the subjects were randomized to diet instruction with two years of follow-up and half to six months of no intervention followed by the same diet instruction and followup. Control subjects had a fasting blood drawn at three months of the nonintervention period. Having parallel intervention and control groups was necessary to test the efficacy of the NCEP Step Two Diet: The diet was taught to study subjects during eight weekly two hour classes. Follow-up included four individual visits, at three, six, nine, and twelve months, with a dietitian and two group sessions, at 4.5 and 10.5 months, in the first year and two individual visits, at 18 and 24 months, in the second year. Fasting blood samples for lipoprotein lipid analysis and 4-day food diaries were collected at all individual visits. Additionally, medical history, lifestyle characteristics, vital signs, other adherence measures, behavioral factors related to adherence, and serum nutrients for monitoring nutrient sufficiency were collected. Dietitians provided adherence and dietary modification counseling as necessary to help participants maximize their adherence. The primary questions to be answered were: 1) Did the NCEP Step Two Diet effectively lower plasma lipids in hypercholesterolemic (HC) and combined hyperlipidemic (CHL) women and men over six months? 2) Did HC and CHL women have a different response than HC and CHL men? 3) Was response in women influenced by menstrual status and sex hormone exposure?, and 4) Were the behavioral adaptations to dietary modification different between women and men?

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-04; Study Completion 1996-09

REFERENCES:
- [Background] Retzlaff BM, Walden CE, McNeney WB, Buck BL, McCann BS, Knopp RH. Nutritional intake of women and men on the NCEP Step I and Step II diets. J Am Coll Nutr. 1997 Feb;16(1):52-61. doi: 10.1080/07315724.1997.10718649. PMID 9013434
- [Background] Walden CE, Retzlaff BM, Buck BL, McCann BS, Knopp RH. Lipoprotein lipid response to the National Cholesterol Education Program step II diet by hypercholesterolemic and combined hyperlipidemic women and men. Arterioscler Thromb Vasc Biol. 1997 Feb;17(2):375-82. doi: 10.1161/01.atv.17.2.375. PMID 9081694
- [Background] McCann BS, Bovbjerg VE, Curry SJ, Retzlaff BM, Walden CE, Knopp RH. Predicting participation in a dietary intervention to lower cholesterol among individuals with hyperlipidemia. Health Psychol. 1996 Jan;15(1):61-4. doi: 10.1037//0278-6133.15.1.61. PMID 8788542
- [Background] Retzlaff BM, Dowdy AA, Walden CE, Bovbjerg VE, Knopp RH. The Northwest Lipid Research Clinic Fat Intake Scale: validation and utility. Am J Public Health. 1997 Feb;87(2):181-5. doi: 10.2105/ajph.87.2.181. PMID 9103094